CLINICAL TRIAL: NCT06047483
Title: A Multicenter, Randomized, Single Blind, Positive Drug and Placebo Parallel Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of HRF2105patch in Relieving Pain of Osteoarthritis
Brief Title: A Trial of HRF2105 Patch in Relieving Pain of Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRF2105-201
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Analgesia and Anti-inflammatory of Osteoarthritis
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HRF2105 patch (Experimental)
  Interventions: Drug: HRF2105 patch
- Loxoprofen patch (Active Comparator)
  Interventions: Drug: Loxoprofen patch
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HRF2105 patch — HRF2105 patch ，external use，once a day
  Arms: HRF2105 patch
Drug: Loxoprofen patch — Loxoprofen patch ，external use，once a day
  Arms: Loxoprofen patch
Drug: placebo — placebo ，external use，once a day
  Arms: placebo

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HRF2105patch in relieving pain of Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Male or female
3. Meeting the diagnostic criteria of knee Articular bone osteoarthritis
4. The target knee joint meeting the VAS scoring requirements
5. K-L grading II-III，and the other knee joint grading is not higher than the target side
6. Able to walk without assistance
7. Willing to take contraceptive measures, female non pregnancy or lactation period

Exclusion Criteria:

1. Concomitant bronchial asthma; Previous aspirin induced asthma (non steroidal anti-inflammatory drugs induced asthma)
2. Active or high-risk bleeding diseases such as gastrointestinal ulcers may worsen due to the use of NSAIDs
3. Have a history of myocardial infarction or undergo coronary artery bypass grafting surgery
4. Having serious cardiovascular, cerebrovascular, hematopoietic, metabolic system diseases or malignant tumors, as determined by the researcher, it is not suitable to participate in this study
5. The combination of mental illnesses such as depression, dementia, and schizophrenia has been determined by researchers to affect the efficacy evaluation of study drugs
6. Arthritis caused by other factors such as dermatomyositis, gouty arthritis, psoriatic arthritis, ankylosing spondylitis, rheumatoid arthritis, purulent arthritis, systemic lupus erythematosus
7. In addition to the knee joint, complications such as goose foot bursitis, intermittent claudication, and other conditions that can cause pain in the knee joint area
8. Severe osteoarthritis with obvious narrowing of joint space and indications for surgery
9. Pain in other areas that affect the evaluation of bone and joint pain, such as hip joint pain or lower back pain
10. Rashes and skin damage on the intended application of the study drug
11. Abnormal liver and kidney function, anemia or thrombocytopenia
12. Within one year prior to signing the ICF, either side of the knee joint experienced open knee injury or underwent other knee joint surgeries such as arthroscopy, arthroscopic debridement, knee replacement, etc
13. Patients who have received intra-articular drug injection therapy (such as glucocorticoids, sodium hyaluronate, medical chitosan, growth factors, and platelet rich plasma) on either side of the knee joint within 3 months prior to signing the ICF
14. Within the first 5 days of randomization or during the study period, other drugs for treating osteoarthritis need to be used except the study drug
15. During the research process, physical therapy and rehabilitation therapy for the lower limbs or waist are required
16. Individuals with a history of allergies or contraindications to any component of this product or other losoprofen sodium preparations
17. During this period, alcohol, drugs, and drug withdrawal may affect the effectiveness and safety evaluation of the study drug
18. Participants in other clinical trials within 3 months
19. Family members of the subjects in this study (cohabiting)
20. Clinical research center employees directly involved in the operation, management, or support of this trial, or immediate family members
21. Other situations that the researcher determines are not suitable for participating in this clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in VAS score from baseline at the end of treatment Day7 on rising from the chair | Day7

SECONDARY OUTCOMES:
Change in WOMAC pain score from baseline at the end of treatment (Day7) | Day7
Change in WOMAC stiffness score from baseline at the end of treatment (Day7) | Day7
Change in WOMAC daily activity score from baseline at the end of treatment (Day7) | Day7
Change in WOMAC total score from baseline at the end of treatment (Day7) | Day7
Daily average dose of remedial drug (Paracetamol) during the treatment period | Day0-Day7
Researcher satisfaction score | Day7
Subject satisfaction score | Day7
Skin irritation and sensitization scores | Day0-Day7

IPD SHARING:
Plan to Share IPD: Undecided